CLINICAL TRIAL: NCT05949307
Title: The Efficacy of Acupuncture and Laser Acupuncture in Treating Chemotherapy or Target Therapy-induced Hand-foot Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Chief and Attending Physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH112-REC1-020
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hand-Foot Syndrome
Keywords: acupuncture; laser acupuncture; chemotherapy; target therapy; hand-foot syndrome
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture group (Experimental): receive acupuncture treatment
  Interventions: Device: acupuncture
- Laser acupuncture group (Experimental): receive laser acupuncture treatment
  Interventions: Device: laser acupuncture
- Sham laser acupuncture group (Sham Comparator): receive sham-laser acupuncture treatment
  Interventions: Device: Sham-laser acupuncture

INTERVENTIONS:
Device: acupuncture — acupuncture
  Arms: Acupuncture group
Device: laser acupuncture — laser acupuncture
  Arms: Laser acupuncture group
Device: Sham-laser acupuncture — Sham-laser acupuncture
  Arms: Sham laser acupuncture group

SUMMARY:
Chemotherapy or target therapy-induced hand-foot syndrome in cancer patients affects the quality of life. At present, there is no better treatment for this side effect of chemotherapy or target therapy. In severe cases, it is necessary to reduce the dose of chemotherapy or target therapy, which may affect the progress and effect of chemotherapy. In recent years, acupuncture has been widely used for many side effects of chemotherapy, such as numbness of hands and feet, gastrointestinal discomfort, and dizziness. There have been many studies have proved to be effective, but quite few studies explored the acupuncture treatment improves the hand-foot syndrome caused by chemotherapy or target therapy in cancer patients. Therefore, the investigators expect to evaluate the efficacy of acupuncture, and applying acupuncture or laser acupuncture to improve hand-foot syndrome caused by chemotherapy or target therapy in cancer patients in the future.

DETAILED DESCRIPTION:
The investigators design a single-center, sham-controlled, assessor- and subject- blind, randomized clinical trial. 60 subjects will be equally and randomly divided into an acupuncture group, laser acupuncture, and sham-laser acupuncture groups in the 6-week trial. Each subject receives acupuncture, laser acupuncture, or sham-laser acupuncture three times a week for three consecutive weeks depending on their group, with a total of 9 times interventions. Outcome measures include Common adverse events evaluation standard version 5.0 (CTCAE) and Visual Analogue Scale (VAS), Dermatology Life Quality Index (DLQI) and assessment of cancer patients' quality of life questionnaire (EORTC QLQ-C30). ANSWatch and Thermal Image Camera are also used to assess those subjects. Those outcome measures will be conducted at baseline, the 3rd and the 6th week after the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients receiving chemotherapy or targeted therapy
2. Age over 20 years old
3. Western medicine diagnoses hand-foot syndrome
4. Sign the consent form

Exclusion Criteria:

1. Pregnant or planning to become pregnant
2. Serious arrhythmia (or cardiac pacemaker installed)
3. Epilepsy
4. Severe organ failure, such as heart and lung failure, liver and kidney failure
5. Psychiatric history, unable to cooperate with acupuncture and assessors
6. Those who received traditional Chinese medicine treatment for hand-foot skin reaction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
The change of Common Terminology Criteria for Adverse Events (CTCAE) version 5. 0 | Change from Baseline severity of hand-foot syndrome at 3 weeks
  Evaluate skin symptoms assessed by Common Terminology Criteria for Adverse Events version 5. 0 (total three grade. Grade 1 is minimal skin changes, and grade 3 is severe skin changes)
The change of scores of Visual analogue scale (VAS) | Change from Baseline severity of pain at 3 weeks
  pain evaluation assessed by Visual analogue scale, score from 0 (no pain) to 10 (unbearable pain)
The change of Dermatology Life Quality Index (questionnaire) | Change from Baseline quality of life at 3 weeks
  evaluate quality of life assessed by Dermatology Life Quality Index
The change of EORTC QLQ-C30 (questionnaire) | Change from Baseline quality of life at 3 weeks
  evaluate quality of life assessed by EORTC QLQ-C30
The change of LF/HF before and after treatment | Change from Baseline LF/HF at 3 weeks
  testing LF/HF assessed by ANSWatch wrist monitor
The change of temperature of limbs before and after treatment | Change from Baseline temperature at 3 weeks
  testing temperature assessed by Thermal Imaging Analysis

SECONDARY OUTCOMES:
The change of Common Terminology Criteria for Adverse Events (CTCAE) version 5. 0 | Change from Baseline severity of hand-foot syndrome at 6 weeks
  Evaluate skin symptoms assessed by Common Terminology Criteria for Adverse Events version 5. 0 (total three grade. Grade 1 is minimal skin changes, and grade 3 is severe skin changes)
The change of scores of Visual analogue scale (VAS) | Change from Baseline severity of pain at 6 weeks
  pain evaluation assessed by Visual analogue scale, score from 0 (no pain) to 10 (unbearable pain)
The change of Dermatology Life Quality Index (questionnaire) | Change from Baseline quality of life at 6 weeks
  evaluate quality of life assessed by Dermatology Life Quality Index
The change of EORTC QLQ-C30 (questionnaire) | Change from Baseline quality of life at 6 weeks
  evaluate quality of life assessed by EORTC QLQ-C30
The change of LF/HF before and after treatment | Change from Baseline LF/HF at 6 weeks
  testing LF/HF assessed by ANSWatch wrist monitorng LF/HF
The change of temperature of limbs before and after treatment | Change from Baseline temperature at 6 weeks
  testing temperature assessed by Thermal Imaging Analysis

IPD SHARING:
Plan to Share IPD: Undecided